CLINICAL TRIAL: NCT00004924
Title: Phase II Trial of Irinotecan Plus Paclitaxel in Patients With Advanced Nonsmall Cell Lung Cancer
Brief Title: Paclitaxel and Irinotecan in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067608; YALE-HIC-10740; NCI-G00-1701
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with irinotecan works in treating patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity and toxicities of irinotecan and paclitaxel in patients with advanced non-small cell lung cancer.

OUTLINE: Patients receive paclitaxel IV over 1 hour followed immediately by irinotecan IV over 30 minutes. Treatment continues weekly for 2 weeks followed by one week of rest. Courses are repeated every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 11-22 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic non-small cell lung cancer for which no curative therapy exists
* Stage IIIB with pleural effusion allowed
* Measurable or evaluable disease
* CNS metastases allowed if disease stable at least 4 weeks following completion of surgery and/or radiotherapy and no anticonvulsant required

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if tumor involves liver)

Renal:

* Creatinine clearance at least 70 mL/min

Other:

* No other malignancies within past 3 years except nonmelanomatous skin cancer and carcinoma in situ of the cervix
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective birth control
* No active infection
* No concurrent medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy for lung cancer
* No prior irinotecan or paclitaxel

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior wide field radiotherapy
* No prior radiotherapy to greater than 20% of bone marrow allowed

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1999-03; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Murren, MD, Study Chair — Yale University
Locations (2):
- United States (2):
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Northwestern Connecticut Oncology-Hematology Associates - Torrington, Torrington, Connecticut